CLINICAL TRIAL: NCT05328050
Title: Local Registry for Data Collection of Patients With Achondroplasia / Hypochondroplasia for Epidemiological, Care and Research Studies
Brief Title: Registry for Patients With Achondroplasia / Hypochondroplasia (OMPR-Ach/Hy)
Acronym: OMPR-Ach/Hy
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Maria Francesca Bedeschi, Principal investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: NaturalhistoryAch2021
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Achondroplasia; Hypochondroplasia
MeSH Terms: conditions — Achondroplasia; Hypochondroplasia | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Achondroplasia
  Interventions: Other: Registry
- Hypochondroplasia
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — observational, data collection

SUMMARY:
This registry is a observational, single-center study designed to collect clinical data on patients with achondroplasia and hypochondroplasia.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of achondroplasia/hypochondroplasia
* Patients (and/or Parents legal guardian when required) able to provide informed consent

Exclusion Criteria:

* Absence of diagnosis of achondroplasia/hypochondroplasia
* Patients (and/or Parents legal guardian when required) not able to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Achondroplasia / Hypochondroplasia afferent to IRCCS Ca' Granda Ospedale Maggiore Policlinico Milano
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Registry of Achondroplasia and Hypochondroplasia Patients | 10 years
  Collection of medical information of achondroplasia and hypochndroplasia patients intended for use in future research studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Genetics Unit, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Milan, Milan, Italy